CLINICAL TRIAL: NCT00529451
Title: An Eight Week, Double-blind, Randomized, Multicenter, Parallel Group, Active-controlled Study Comparing the Safety and Efficacy of Aliskiren 300 mg, 150 mg and 75 mg to Ramipril 5 mg in Patients With Essential Hypertension
Brief Title: Safety and Efficacy of Aliskiren 300 mg, 150 mg and 75 mg in Patients With Essential Hypertension Compared to Ramipril 5 mg
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: External Affairs, Novartis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CSPP100A2339
Record Dates: First submitted 2007-09-12; First posted 2007-09-14 (Estimated); Results first posted 2011-03-25 (Estimated); Last update posted 2011-03-25 (Estimated); Status verified 2011-02

CONDITIONS: Hypertension
Keywords: Hypertension, Aliskiren, Ramipril
MeSH Terms: conditions — Hypertension | interventions — aliskiren; Ramipril

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Aliskiren 300 mg (Experimental): Aliskiren 300 mg once daily
  Interventions: Drug: Aliskiren
- Aliskiren 150 mg (Experimental): Aliskiren 150 mg once daily
  Interventions: Drug: Aliskiren
- Aliskiren 75 mg (Experimental): Aliskiren 75 mg once daily
  Interventions: Drug: Aliskiren
- Ramipril 5 mg (Active Comparator): Ramipril 5 mg once daily
  Interventions: Drug: Ramipril

INTERVENTIONS:
Drug: Aliskiren — Aliskiren
  Arms: Aliskiren 150 mg; Aliskiren 300 mg; Aliskiren 75 mg
Drug: Ramipril — comparator
  Arms: Ramipril 5 mg

SUMMARY:
This study is designed to investigate the efficacy, safety and tolerability of aliskiren 300 mg, 150 mg and 75 mg when compared to ramipril 5 mg in patients with essential hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have msDBP ≥ 90 mmHg and < 110 mmHg at the visit immediately prior to Visit 3
* Patients must have msDBP >OR= 95 mmHg and < 110 mmHg at Visit 3
* Patients must have an absolute difference of < or =10 mmHg in their mean sitting diastolic blood pressure (msDBP) from Visit 2 to Visit 3

Exclusion Criteria:

* Severe hypertension (grade 3 WHO classification; msDBP >or= 110 mmHg and/or msSBP >or = 180 mmHg).
* History or evidence of a secondary form of hypertension.
* History of transient ischemic cerebral attack within 12 months of visit 1.
* Current angina pectoris requiring pharmacological therapy (other than those patients on a stable dose of oral or topical nitrates)
* Type 1 or Type 2 diabetes mellitus with glycosylated hemoglobin (HbA1c) > 8% at Visit 1.
* Known or suspected contraindications to the study medications, including history of allergy to ramipril or other ACE Inhibitors.

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1613 (Actual)
Dates: Start 2007-09; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Chair — Novartis
Locations (3):
- Novartis Investigative Sites, China, China
- Novartis Investigative Sites, India, India
- Novartis Investigative Sites, Thailand, Thailand

REFERENCES:
- [Derived] Wang GM, Li LJ, Tang WL, Wright JM. Renin inhibitors versus angiotensin converting enzyme (ACE) inhibitors for primary hypertension. Cochrane Database Syst Rev. 2020 Oct 22;10(10):CD012569. doi: 10.1002/14651858.CD012569.pub2. PMID 33089502

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Aliskiren 300 mg | Aliskiren 150 mg | Aliskiren 75 mg | Ramipril 5 mg
Started | 331 | 323 | 332 | 330
Completed | 294 | 275 | 292 | 299
Not Completed | 37 | 48 | 40 | 31
Not completed — Subject withdrew consent | 16 | 21 | 13 | 12
Not completed — Adverse Event | 9 | 16 | 14 | 8
Not completed — Unsatisfactory therapeutic response | 6 | 2 | 5 | 4
Not completed — Lost to Follow-up | 4 | 7 | 4 | 4
Not completed — Protocol deviation | 1 | 1 | 4 | 1
Not completed — Administrative problems | 1 | 1 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aliskiren 300 mg | Aliskiren 150 mg | Aliskiren 75 mg | Ramipril 5 mg | Total
Number analyzed (Participants) | 331 | 323 | 332 | 330 | 1316
Age Continuous [Mean (Standard Deviation); unit: years] | 53.8 (9.45) | 53.3 (10.53) | 52.7 (10.22) | 52.9 (9.60) | 53.2 (9.95)
Age, Customized [Number; unit: Participants]
  < 65 years | 288 | 273 | 285 | 296 | 1142
  ≥ 65 years | 43 | 50 | 47 | 34 | 174
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 150 | 140 | 144 | 151 | 585
  Male | 181 | 183 | 188 | 179 | 731

OUTCOME MEASURES:

1. Secondary Outcome: Change in Mean Sitting Systolic Blood Pressure (msSBP)and Mean Sitting Diastolic Blood Pressure (msDBP) From Baseline to 8 Week Endpoint
Description: To evaluate the change in Mean Sitting Systolic Blood Pressure (msSBP) and Mean Sitting Diastolic blood Pressure (msDBP) from baseline to 8 week endpoint on aliskiren 300 mg, 150 mg and 75 mg vs. ramipril 5 mg in patients with essential hypertension.
Time Frame: Baseline and Week 8
Population: Intent-to-treat. Analyzed patients received at least one dose of study drug and had a post baseline measurement.
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Aliskiren 300 mg | Aliskiren 150 mg | Aliskiren 75 mg | Ramipril 5 mg
Number analyzed (Participants) | 327 | 318 | 324 | 323
mm Hg
  msSBP | -14.39 (0.66) | -12.16 (0.67) | -12.24 (0.66) | -11.46 (0.66)
  msDBP | -11.63 (0.44) | -10.04 (0.44) | -10.66 (0.44) | -9.19 (0.44)

2. Secondary Outcome: Evaluation of the Percentage of Patients Controlled to a Target Blood Pressure of < 140/90 mmHg on Aliskiren 300 mg, 150 mg and 75 mg vs. Ramipril 5 mg
Description: To evaluate the percentage of patients controlled to a target blood pressure of < 140/90 mmHg on aliskiren 300 mg, 150 mg and 75 mg vs. ramipril 5 mg.
Time Frame: Week 8
Population: Intent-to-treat. Analyzed patients received at least one dose of study drug and had a post baseline measurement.
Measure: Number; unit: Percentage of participants
Arm/Group | Aliskiren 300 mg | Aliskiren 150 mg | Aliskiren 75 mg | Ramipril 5 mg
Number analyzed (Participants) | 327 | 318 | 324 | 323
Percentage of participants | 52.29 | 48.11 | 45.68 | 43.65

3. Secondary Outcome: Evaluation of the Percentage of Responders on Aliskiren 300 mg, 150 mg and 75 mg vs. Ramipril 5 mg, Define as msDBP < 90 mmHg or ≥ 10mmHg Decrease From Baseline in msDBP
Description: To evaluate the percentage of responders on aliskiren 300 mg, 150 mg and 75 mg vs. ramipril 5 mg, defined as msDBP < 90 mmHg or ≥ 10mmHg decrease from baseline in msDBP.
Time Frame: Week 8
Population: Intent-to-treat. Analyzed patients received at least one dose of study drug and had a post baseline measurement.
Measure: Number; unit: Percentage of participants
Arm/Group | Aliskiren 300 mg | Aliskiren 150 mg | Aliskiren 75 mg | Ramipril 5 mg
Number analyzed (Participants) | 327 | 318 | 324 | 323
Percentage of participants | 67.89 | 59.75 | 59.57 | 53.87

4. Primary Outcome: Non-inferiority of Aliskiren 300 mg to Ramipril 5 mg in Change in Mean Sitting Diastolic Blood Pressure (msDBP)
Description: To evaluate the non-inferiority of aliskiren 300 mg to ramipril 5 mg in the change in Mean Sitting Diastolic Blood Pressure (msDBP) from baseline to 8 week endpoint
Time Frame: Baseline and Week 8
Population: Intent-to-treat. Analyzed patients received at least one dose of study drug and had a post baseline measurement.
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Aliskiren 300 mg | Ramipril 5 mg
Number analyzed (Participants) | 327 | 323
mm Hg | -11.63 (0.44) | -9.19 (0.44)
Statistical Analysis 1: Comparison: Aliskiren 300 mg vs Ramipril 5 mg; Test type: Non-Inferiority or Equivalence — Non-inferiority margin of 2.25 mm Hg; Mean Difference (Final Values) = -2.44, 95% CI 2-sided [-3.63 to -1.25]

5. Primary Outcome: Non-inferiority of Aliskiren 150 mg to Ramipril 5 mg in Change in Mean Sitting Diastolic Blood Pressure (msDBP)
Description: as for outcome 4
Time Frame: Baseline and Week 8
Population: Intent-to-treat. Analyzed patients received at least one dose of study drug and had a post baseline measurement.
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Aliskiren 150 mg | Ramipril 5 mg
Number analyzed (Participants) | 318 | 323
mm Hg | -10.04 (0.44) | -9.19 (0.44)
Statistical Analysis 1: Comparison: Aliskiren 150 mg vs Ramipril 5 mg; Test type: Non-Inferiority or Equivalence — Non-inferiority margin of 2.25 mm Hg; Mean Difference (Final Values) = -0.86, 95% CI 2-sided [-2.06 to 0.34]

6. Primary Outcome: Non-inferiority of Aliskiren 75 mg to Ramipril 5 mg in Change in Mean Sitting Diastolic Blood Pressure (msDBP)
Description: To evaluate the non-inferiority of aliskiren 75 mg to ramipril 5 mg in the change in Mean Sitting Diastolic Blood Pressure (msDBP) from baseline to 8 week endpoint
Time Frame: Baseline and Week 8
Population: Intent-to-treat. Analyzed patients received at least one dose of study drug and had a post baseline measurement.
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Aliskiren 75 mg | Ramipril 5 mg
Number analyzed (Participants) | 324 | 323
mm Hg | -10.66 (0.44) | -9.19 (0.44)
Statistical Analysis 1: Comparison: Aliskiren 75 mg vs Ramipril 5 mg; Test type: Non-Inferiority or Equivalence — Non-inferiority margin of 2.25 mm Hg; Mean Difference (Final Values) = -1.48, 95% CI 2-sided [-2.67 to -0.28]

ADVERSE EVENTS:
Time Frame: 8 weeks
Description: One randomized patient in the Ramipril group never received blinded study medication. The subject is therefore not included in the "at risk" population.
Arm/Group | Aliskiren 300 mg | Aliskiren 150 mg | Aliskiren 75 mg | Ramipril 5 mg
Serious Adverse Events (participants affected / at risk) | 1/331 | 2/323 | 3/332 | 1/329
Other Adverse Events (participants affected / at risk) | 4/331 | 3/323 | 2/332 | 17/329
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Aliskiren 300 mg (N=331) | Aliskiren 150 mg (N=323) | Aliskiren 75 mg (N=332) | Ramipril 5 mg (N=329)
Chest pain (General disorders) | 0 | 0 | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Medical device complication (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 1 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1
Varicose vein (Vascular disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Aliskiren 300 mg (N=331) | Aliskiren 150 mg (N=323) | Aliskiren 75 mg (N=332) | Ramipril 5 mg (N=329)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 3 | 2 | 17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.